CLINICAL TRIAL: NCT06163469
Title: Instillation in Neurogenic Bladders to Decrease Unplanned Healthcare Encounters
Brief Title: Effect of Chlorhexidine Gluconate Bladder Instillations in Patients With Chronic Suprapubic Catheters on Unplanned Healthcare Encounters and Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Irrimax Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000034836; 000 (Other: CTGTY)
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Neurogenic Bladder; Urinary Retention
Keywords: recurrent UTI; bladder irrigation
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Urinary Retention; Urinary Tract Infections | interventions — Administration, Intravesical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Arm I (Experimental): Participants will get bladder instillations of normal saline for three months and then six months of instillations with chlorohexidine gluconate. After the instillation phase the patients will undergo an observational phase with six months of catheter exchanges without the intervention.
  Interventions: Device: Bladder instillation with Irrisept

INTERVENTIONS:
Device: Bladder instillation with Irrisept — 9 months of bladder instillations (3 months of saline and 6 months of chlorohexidine gluconate)

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility and tolerability of 0.05% Chlorhexidine Gluconate (CGH) bladder instillations in an outpatient setting at the time of suprapubic catheter (SPC) exchange in patients with history of recurrent urinary tract infections (UTI). The main questions are:

1. is instillation of 150mL of CGH for five-minute duration at the time of SPC exchange feasible in an outpatient setting and tolerable for patients.
2. does this protocol decrease the rate of unplanned health care visits and improve patient quality of life.

Patients will undergo the treatment protocol during their routine suprapubic catheter exchanges.

DETAILED DESCRIPTION:
Bacterial colonization is present in up to 95% of chronically catheterized patients. Although a positive urine culture collected from an indwelling catheter is not in isolation indicative of an acute urinary tract infection (UTI), long term catheter use is associated with increased rates of recurrent urinary tract infections (rUTI), pyelonephritis, and bacteremia. Using antibiotics for prevention of infections in this patient population can be challenging given the side effects, cost, and emergence of resistant bacteria with antibiotic therapy. To limit systemic side effects, intravesical irrigation is a promising route of medication administration. The use of a non-antibiotic anti-microbial at the time of SPC exchange would eliminate the obstacles of non-compliance and antibiotic resistance associated with antibiotic irrigation for preventive therapy. Irrisept, a 0.05% Chlorhexidine Gluconate (CHG) irrigation in sterile water, could be a promising agent to reduce symptomatic UTIs and unplanned tube changes in chronically catheterized patients.

The proposed route of intravesical instillation involves the administration of a therapeutic agent directly into the bladder via a urinary catheter. This route allows for local contact with bladder mucosa and urinary pathogens. It is a currently accepted route of administration used for therapeutics in urologic conditions including, but not limited to UTI prophylaxis, bladder cancer, hemorrhagic cystitis, and interstitial cystitis. Benefits of intravesical instillation include maximizing exposure of the therapeutic within the bladder while limiting systemic absorption and side effects.

A volume 150cc is based on current clinical administration of bladder instillations. Current intravesical drug delivery is most commonly utilized in volumes 50-150cc for in-office instillation. Population studies of normal volunteers demonstrate that 1st bladder sensation occurs between 125-200cc with subsequent desire to void occurring between 170-370cc. Increasing instillation volumes greater than 150cc, especially in the chronically catheterized population, can lead to patient discomfort or dysreflexia and inability to tolerate the therapy without analgesia or anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Indwelling suprapubic catheter with insertion date at least 1 year prior to study enrollment date.
* History of urinary tract infections, treated for at least 1 positive urine culture in last 6 months

Exclusion Criteria:

* Current radiographic evidence of urolithiasis
* History of vesicoureteral reflux
* History of renal transplantation
* History of bladder augmentation
* Inability to stop use of other rUTI prophylaxis treatments for the duration of their trial enrollment
* Life expectancy of less than 12 months prior to consent.
* Known hypersensitivity or allergy to chlorhexidine.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
tolerability and feasibility of CGH bladder instillation | 9 months
  Tolerability and feasibility of CGH bladder instillation of 150mL for five-minute duration at the time of SPC exchange. Volumes of each instillation and tolerated dwell time will be recorded with each instillation.

SECONDARY OUTCOMES:
Incidence of bacteriuria | monthly for 15 months
  Urine cultures will be taken at each SPC exchange for nine months while undergoing irrigations (3 months with saline and 6 months with Irrisept) and for an additional six months following completion of instillation treatment. Incidence of bacteriuria prior to the start of instillation will be compared to the incidence during the instillation phase and observation phase.
effect of chlorhexidine gluconate catheter biofilm flora | up to 9 months
  the catheter tips will be sent for culture at each exchange. results between the saline and CGH irrigations will be compared
Incidence of symptomatic UTI | up to 15 months
  Participants will complete a validated UTI symptom assessment at the time of instillation and then three days later when the urine culture is finalized. Responses will be compared to each participants self reported typical UTI symptoms to differentiate between asymptomatic bacteruria and symptomatic UTI.
impact of mechanical bladder washing | up to 9 months
  Urine culture results and patient questionnaires during the saline irrigations will be compared to those during the CGH irrigation
effect of chlorhexidine changes the microbiome of the bladder | up to 15 months
  Urine culture data from the CGH instillation phase will be compared to culture data from the saline irrigation and observational period. Changes in the dominant bacteria from each culture will be reported.
unplanned healthcare contact between routine SPC exchanges | up to 15 months
  At each SPC change and instillation an interval history will be taken any unplanned healthcare utilization (I.e. emergency room, primary care, and urology calls and visits) will be recorded. The number of recorded events during the instillation and observation phases will be compared.
patient quality of life and overall satisfaction | up to 15 months
  participants will complete a validated six question quality of life questionnaire at months 0, 3, 6, 9, 12, and 15. Changes in the sum total (lower the sum the higher the quality of life) and individual responses will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Sterling, MD, MSc, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Health, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal.